CLINICAL TRIAL: NCT00781534
Title: A Clinical Trial of Ginseng for Glucose Intolerance
Brief Title: A Clinical Trial of Ginseng in Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Kenneth S. Polonsky, MD, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 03-0824
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Diabetes
Keywords: Health Supplements; Ginseng; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Asian ginseng; ginsenoside Re; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. Ginseng (Active Comparator): Ginseng group
  Interventions: Drug: Ginseng
- 2. Ginsenosdie RE (Active Comparator): Ginsenoside RE (a metabolite of ginseng) group
  Interventions: Drug: Ginseng; Drug: ginsenoside RE
- 3. Placebo (Placebo Comparator): placebo ("sugar" pill) group
  Interventions: Dietary Supplement: Placebo (sugar pill)

INTERVENTIONS:
Drug: Ginseng — Each of the 3 arms will be compared to determine if there is any clinical difference in blood sugars between the 3 groups
  Arms: 1. Ginseng
Drug: Ginseng
  Arms: 2. Ginsenosdie RE
Drug: ginsenoside RE — active metabolite of ginseng
  Arms: 2. Ginsenosdie RE
Dietary Supplement: Placebo (sugar pill) — placebo group
  Arms: 3. Placebo

SUMMARY:
a clinical study of Ginseng its potential affect on diabetes

DETAILED DESCRIPTION:
Comparing three groups (those with & without normal blood sugar levels) to see if there is any clinically significant change in blood sugar levels in relationship to those taking:

1. ginseng
2. ginsenoside RE (a type of metabolized ginseng)
3. placebo

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65
* healthy, non-diabetic
* healthy, impaired glucose tolerance/mild diabetes (no medications required)

Exclusion Criteria:

* impaired glucose tolerance (borderline diabetes that requires medications)
* diabetes (requiring medications)
* caffeine sensitivity
* known cardiac, peripheral vascular diseases
* arrhythmias (irregular heart rhythms)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-09; Primary Completion 2004-12 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Polonsky, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Reeds DN, Patterson BW, Okunade A, Holloszy JO, Polonsky KS, Klein S. Ginseng and ginsenoside Re do not improve beta-cell function or insulin sensitivity in overweight and obese subjects with impaired glucose tolerance or diabetes. Diabetes Care. 2011 May;34(5):1071-6. doi: 10.2337/dc10-2299. Epub 2011 Mar 16. PMID 21411505